CLINICAL TRIAL: NCT07000903
Title: Occupational and Environmental Causes of Autoimmune Diseases: Clarifying Epidemiology and Improving Detection
Brief Title: Occupational and Environmental Causes of Autoimmune Diseases
Acronym: EXIMIOUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021/21SEP/388
Record Dates: First submitted 2022-06-20; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Lupus Erythematosus, Systemic; Systemic Sclerosis; Rheumatoid Arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Verify the added value of environmental exposure and immunophenotyping to establish a possible etiology of AID: the exposure and immune profiles will be determined in HBM blood and urine samples collected prospectively during the first SOC visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure and immune profiles (Experimental): The exposure and immune profiles will be determined in HBM blood and urine samples collected prospectively during the first SOC visit.
  Interventions: Other: Exposure and immune profiles

INTERVENTIONS:
Other: Exposure and immune profiles — The exposure and immune profiles will be determined in HBM blood and urine samples collected prospectively during the first SOC visit.

SUMMARY:
The investigators hypothesize that part of the systemic autoimmune diseases (AID) patients might prove to have an occupational or environmental disease which is potentially preventable. The recognition of the occupational or environmental etiology of autoimmune disorders has major implications for patients and society and will generate opportunity for prevention and meaningful clinical intervention. The investigators intend to use the urine/blood exposure measurements to demonstrate the etiological role of environment in patients developing AID patients.

The investigators are mounting an epidemiological study to elucidate the environmental etiology of AID and their effects on the immune profile and disease course. A population-based case-control study will be done with adult patients with newly diagnosed systemic sclerosis, systemic lupus erythematosus, rheumatoid arthritis (n=100 per disease).

DETAILED DESCRIPTION:
Systemic autoimmune diseases (AID) regroup a broad range of related diseases characterized by self-damaging immune responses. They mainly comprise systemic lupus, systemic sclerosis and rheumatoid arthritis and remain a significant clinical challenge. Rheumatoid arthritis (RA) is a degenerative disease associated with chronic inflammation that ultimately leads to joint damage, deformation and destruction. Systemic lupus erythematosus (SLE) is characterized by tissue injury resulting from immune responses and serological changes. This multifaceted etiology AID is initiated by the loss of tolerance to self-antigens and the accumulation of autoreactive B and T cells that promote autoreactive antibody production, immune complex formation and activated mononuclear cell infiltration in affected tissues. Finally, small vessels-vasculopathology, internal tissue fibrogenesis and thickening skin characterize systematic sclerosis (SSc) patients. These lesions derive from dysregulated immune functions altering connective tissue integrity.

Several risk factors have been pinpointed to explain the triggering of these AID. Scientists have managed to identify the main genetic factors. Susceptibility to AID is strongly associated to MHC class II polymorphisms and adaptive immunity activation (particularly effector T lymphocytes).

Nevertheless, several studies have also emphasized the contribution of environmental factors, which may function as triggers of innate immunity and may contribute to the breakdown of self-tolerance by modifying protein antigens. Cigarette smoking has proven to be a strong risk factor for seropositive RA and SLE. Cigarette smoke leads to post-translational modifications of antigens by citrullination (citrullinated antigens) that induce the production of anticitrullinated protein antibodies (ACPA) and the onset of ACPA-positive RA. Occupational factors may also cause or trigger AID. In a retrospective study conjointly performed by the Cliniques Universitaires Saint-Luc (CUSL) and UZ Leuven, it was concluded that an estimated 50% of male patients suffering from SSc have occupational exposure to silica and solvents. These findings indicate that environmental factors can provide clinically useful information in the management of AID patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically active lupus; systemic sclerosis; rheumatoid arthritis
* At least 18 years old
* Without first line disease-modifying therapy
* Written informed consent must be obtained before any assessment is performed

Exclusion Criteria:

* Younger than 18
* Wearers of metal prostheses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Exposome: quantification of the exposure of patients to environmental agents | Through the entire study, approximately during 30 months
  exposure to different environmental pollutants is different in cases with systemic lupus erythematosus, systemic sclerosis, and rheumatoid arthritis.
Exposome: quantification of the exposure of patients to agents | Through the entire study, approximately during 30 months
  exposure to different occupational pollutants is different in cases with systemic lupus erythematosus, systemic sclerosis, and rheumatoid arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: François Huaux, Pr, Study Director — UCLouvain - IREC
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium